CLINICAL TRIAL: NCT04228978
Title: PROmote Weight Loss in Obese Peripheral Artery Disease (PAD) Patients to preVEnt Mobility Loss: The PROVE Trial
Brief Title: Promote Weight Loss in Obese Peripheral Artery Disease (PAD) Patients to Prevent Mobility Loss
Acronym: PROVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Wake Forest University (Other)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00209524; UG3HL141729-01A1 (NIH)
Record Dates: First submitted 2019-12-08; First posted 2020-01-14 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Artery Disease; Overweight or Obesity
MeSH Terms: conditions — Peripheral Arterial Disease; Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors performing outcome measures will be unaware of participants' group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight loss + exercise (WL+EX) (Experimental): Weight loss + home based walking exercise (WL+EX)
  Interventions: Behavioral: Weight loss; Behavioral: Exercise
- Exercise alone (EX) (Active Comparator): Home based walking exercise (EX)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Weight loss — Walking exercise combined with weight loss
  Arms: Weight loss + exercise (WL+EX)
Behavioral: Exercise — Walking exercise

SUMMARY:
The PROVE Trial is a randomized clinical trial that will determine whether a weight loss intervention combined with walking exercise achieves greater improvement or less decline in six-minute walk distance at 12 month follow-up than walking exercise alone in people with PAD and BMI>25 kg/m2. The intervention uses a Group Mediated Cognitive Behavioral framework, connective mobile technology, remote monitoring by a coach, and a calorie restricted Dietary Approaches to Stop Hypertension (DASH)-derived Optimal Macronutrient Intake Trial for Heart Health (OMNIHeart) diet.

212 participants with PAD and BMI > 25 kg/m2 will be randomized to one of two groups: weight loss + exercise (WL+EX) vs. exercise alone (EX). Participants will be randomized at Northwestern, Tulane University, and University of Minnesota. Our primary outcome is change in six-minute walk distance at 12-month follow-up. Secondary outcomes are change in 6-minute walk distance at 6-month follow-up and change in exercise adherence, physical activity, patient-reported walking ability (measured by the Walking Impairment Questionnaire (WIQ) distance score), and mobility (measured by the Patient-Reported Outcomes Measurement Information System [PROMIS] mobility questionnaire) at 12-month follow-up. Tertiary outcomes are perceived exertional effort (measured by the Borg scale at the end of the 6-minute walk at 12-month follow-up), and diet quality. Exploratory outcomes consist of change in the short physical performance battery (SPPB), the WIQ stair climbing and walking speed scores, and calf muscle biopsy measures at 12-month follow-up. Study investigators will perform calf muscle biopsies in 50 participants to compare changes in mitochondrial biogenesis and activity, capillary density, and inflammation between WL+EX vs. EX.

ELIGIBILITY:
Inclusion criteria are a) presence of PAD; b) BMI> 25 kg/m2; c) Age >= 18. The diagnosis of PAD will be based on the following. First, an ankle brachial index (ABI) value <= 0.90, which is a well-accepted standard for diagnosing PAD. People with a toe brachial index of <=0.70, performed at the study visit, will be eligible. Second, people with an ABI of >0.90 and <=1.00 who experience a 20% or greater drop in ABI in either leg after the heel-rise test will also be included. Third, potential participants with an ABI > 0.90 who provide vascular laboratory evidence or angiographic evidence of PAD will be included. Prior vascular laboratory evidence consists of objective evidence of PAD including toe brachial index (TBI) < 0.70, Duplex measure showing 70% stenosis or greater, a post-exercise ABI drop in either leg of 20% or greater, or ABI values <= 0.90. Angiographic evidence of PAD consists of a stenosis of 70% or greater in a lower extremity artery. Fourth, people with a history of lower extremity revascularization who do not meet the criterion above and have an ABI > 0.90 with a 20% or higher drop in ABI after an exercise test will be eligible if they have symptomatic PAD. Symptomatic PAD will be defined as leg symptoms associated with exertion that resolved within 10 minutes of rest. The presence of symptomatic PAD will be determined based on the claudication questionnaire, the six-minute walk, or principal investigator interview/discussion with the potential participant. The post-exercise ABI drop will be measured by obtaining an ABI, having the participant exercise, and then immediately repeating the ABI. The exercise may consist of either the six-minute walk test or the heel-rise test. The heel-rise test consists of 50 heel rises at a rate of one per second. From the beginning of the trial until early 2023, we used the BMI inclusion criterion of > 28 kg/m2 because overweight and obesity are defined as a BMI of 25 to 29 kg/m2 and > 30 kg/m2, respectively, and because in our PAD cohorts, those with BMI > 28 kg/m2 have significantly greater functional impairment and faster functional decline than those with BMI of 20-28 kg/m2. In order to increase the rate of recruitment, on 1/19/2022, investigators reduced the BMI inclusion criterion to > 25 kg/ m2. People with BMI above 25 are overweight or obese and therefore are expected to benefit from the healthy lifestyle intervention.

Exclusion Criteria:

1. Above or below knee amputation, critical limb ischemia, or wheelchair confinement.
2. Walking is limited by a condition other than PAD.
3. Failure to complete the study run-in, defined as not entering at least 800 Kcal of consumed calories per day for at least five days during the 14-day run-in*.
4. Major surgery, coronary or leg revascularization in the past 3 months or anticipated in the next year.
5. Experienced a heart attack or stroke in the past 3 months.
6. Major medical illness including lung disease requiring oxygen or life-threatening illness, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent.
7. Mini-Mental Status Examination (MMSE) score < 23, dementia and substance abuse. Potential participants with an MMSE score of less than 23 may be eligible if the principal investigator determines that their lower score is due to reasons other than poor cognition. Other potential reasons for lower scores include poor literacy or that English is not their first language.
8. History of being treated for new onset or an acute episode of schizophrenia or psychosis in the past 6 months.
9. Hospitalization for a psychiatric disorder in the past 6 months.
10. BMI > 45 kg/m2
11. History of a significant eating disorder that has been active within the past 5 years or any weight loss treatment in the past 6 months. Weight loss treatment includes weight watchers, any history of weight loss surgery, and using weight loss medications now or in the past six months.
12. Weight gain or loss of more than 25 pounds in the past six months
13. Potential participants unwilling/unable to use a smart phone and unwilling to attend weekly study sessions.
14. Excessive alcohol use, defined as >14 drinks/week in men and > 10 alcoholic drinks/week in women.
15. Current ulcer on bottom of foot
16. Current participation in supervised treadmill exercise, participation in supervised treadmill exercise in the past three months, or planning to participate in supervised treadmill exercise in the next year
17. Increase in angina or angina at rest. Potential participants may become eligible following an abnormal baseline treadmill stress test if they have evidence of an absence of coronary ischemia based on testing with their own physician.
18. Non-English speaking
19. Visual impairment that limits walking ability
20. Currently walking regularly for exercise at a level comparable to the amount of exercise prescribed in the intervention
21. Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
22. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant

    * The run-in will also be used to assist participants with learning the app. However, they must demonstrate ability to enter at least 800 Kcal per day for at least five days of the run-in.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
12-month change in six-minute walk distance | Baseline to 12 months
  Change in six-minute walk distance at 12-month follow-up will be compared between individuals randomized to weight loss + exercise vs. those randomized to exercise alone.

SECONDARY OUTCOMES:
12-month change in minutes of walking exercise/week | Baseline to 12 months
  Change in minutes walked for exercise in a week will be compared between individuals randomized to the weight loss + exercise vs. those randomized to exercise alone at 12-month follow-up.
12-month change in physical activity measured by accelerometer data | Baseline to 12 months
  Change in physical activity at 12-month follow-up will be compared between individuals randomized to the weight loss + exercise vs. those randomized to exercise alone. Change in physical activity will be compared using accelerometer data.
12-month change in Walking Impairment Questionnaire (WIQ) distance score | Baseline to 12 months
  Change in Walking Impairment Questionnaire (WIQ) distance score at 12-month follow-up will be compared between individuals randomized to the weight loss + exercise vs. those randomized to exercise alone. The WIQ distance score ranges from 0-100 with a higher score indicating a better outcome.
12-month change in Patient-Reported Outcomes Measurement Information System (PROMIS) mobility questionnaire | Baseline to 12 months
  Change in Patient-Reported Outcomes Measurement Information System (PROMIS) mobility questionnaire score at 12-month follow-up will be compared between individuals randomized to the weight loss + exercise vs. those randomized to exercise alone. A higher score is better. There is no set minimum and maximum values for the PROMIS questionnaire. However, a higher PROMIS score indicates a better outcome.
6-month change in 6-minute walk distance | Baseline to 6 months
  Change in six-minute walk distance at 6-month follow-up will be compared between individuals randomized to weight loss + exercise vs. those randomized to exercise alone.

OTHER OUTCOMES:
12-month change in perceived exertional effort at the end of the six-minute walk test | Baseline to 12 months
  Change in perceived exertional effort at the end of the six-minute walk test at 12-month follow-up will be compared between individuals randomized to the weight loss + exercise vs. those randomized to exercise alone. Perceived exertional effort will be measured using the Borg scale. The Borg scale is a 15-point scale ranging from six to 20. A higher score indicates greater perceived exertion.
12-month change in diet quality measured by change in Healthy Eating Index | Baseline to 12 months
  Change in diet quality measured by change in Healthy Eating Index (HEI) will be compared between individuals randomized to weight loss + exercise vs. those randomized to exercise alone. Change in diet quality will be measured at 12-month follow-up. The maximum HEI score is 100 points. A higher total HEI score indicates a diet that aligns better with dietary recommendations.
Change in the short physical performance (SPPB) battery questionnaire at 12-month follow-up | Baseline to 12 months
  Change in the short physical performance (SPPB) battery questionnaire will be compared between individuals randomized to weight loss + exercise vs. those randomized to exercise alone. The SPPB questionnaire ranges from 0 to 12 (12 = best).
Change in the WIQ walking speed score at 12-month follow-up | Baseline to 12 months
  Change in the WIQ walking speed score at 12-month follow-up will be compared between individuals randomized to weight loss + exercise vs. those randomized to exercise alone. The WIQ walking speed score ranges from 0-100. A higher score is better.
12-month change in calf muscle biopsy measured COX enzyme activity | Baseline to 12 months
  In a subset of 50 participants, study investigators will compare improvement in calf muscle biopsy measures of mitochondrial activity (COX enzyme activity) between individuals randomized to weight loss + exercise vs. those randomized to exercise alone.
12-month change in the calf muscle biopsy measure mitochondrial biogenesis (PGC-1α) | Baseline to 12 months
  In a subset of 50 participants, study investigators will compare the calf muscle biopsy measures of mitochondrial biogenesis (PGC-1α) between individuals randomized to weight loss + exercise vs. those randomized to exercise alone.
Change in the WIQ stair climbing questionnaire score at 12-month follow-up | Baseline to 12 months
  Change in the WIQ stair climbing questionnaire score at 12-month follow-up will be compared between individuals randomized to weight loss + exercise vs. those randomized to exercise alone. The WIQ stair climbing score ranges from 0-100. A higher score is better.
12-month change in capillary density (capillaries per muscle fiber) | Baseline to 12 months
  In a subset of 50 participants, study investigators will compare calf muscle biopsy measures of capillary density (capillaries per muscle fiber) between individuals randomized to weight loss + exercise vs. those randomized to exercise alone. Change in capillary density will be measured at 12-month follow-up.
12-month change in calf muscle inflammation (IL-6, TNF-α, and IL1β) | Baseline to 12 months
  In a subset of 50 participants, study investigators will compare calf muscle biopsy measures of calf muscle inflammation (IL-6, TNF-α, and IL1β) between individuals randomized to weight loss + exercise vs. those randomized to exercise alone. Change in calf muscle inflammation will be measured at 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mary M McDermott, MD, Principal Investigator — Northwestern University; Walter Ambrosius, PhD, Principal Investigator — Wake Forest University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whipple MO, Pfammatter AF, Spring B, Rejeski WJ, Treat-Jacobson D, Domanchuk KJ, Dressler EV, Ferrucci L, Gildea L, Guralnik JM, Harvin L, Leeuwenburgh C, Polonsky TS, Reynolds E, Stowe CL, Sufit R, Van Horn L, Walkup MP, Ambrosius WT, McDermott MM. Study Design, Rationale, and Methodology for Promote Weight Loss in Patients With Peripheral Artery Disease Who Also Have Obesity: The PROVE Trial. J Am Heart Assoc. 2023 Sep 5;12(17):e031182. doi: 10.1161/JAHA.123.031182. Epub 2023 Aug 29. PMID 37642035